CLINICAL TRIAL: NCT06373055
Title: Prediction of Therapeutic Response to Neoadjuvant Chemotherapy in Muscle Invasive Bladder Cancer Patients Using Spatial Transcriptomics
Status: Recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2023-1232
Record Dates: First submitted 2023-12-12; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Muscle-invasive Bladder Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Platinum-based Neoadjuvant Chemotherapy Sensitive Patients: Patients with newly confirmed muscle-invasive bladder cancer who have favorable treatment response to platinum-based neoadjuvant chemotherapy
  Interventions: Other: neoadjuvant chemotherapy followed by radical cystectomy
- Platinum-based Neoadjuvant Chemotherapy Resistant Patients: Patients with newly confirmed muscle-invasive bladder cancer who have unfavorable treatment response to platinum-based neoadjuvant chemotherapy
  Interventions: Other: neoadjuvant chemotherapy followed by radical cystectomy

INTERVENTIONS:
Other: neoadjuvant chemotherapy followed by radical cystectomy — combination of dose-dense methotrexate, vinblastine, doxorubicin, and cisplatin (ddMVAC) or combination of gemcitabine and cisplatin (GC) followed by radical cystectomy

SUMMARY:
Although neoadjuvant chemotherapy in muscle-invasive bladder cancer has significantly improved oncological outcomes, approximately 50% of patients do not respond to neoadjuvant chemotherapy, which has adverse effects on patients by causing treatment toxicity and surgical delays. Therefore, treatment tailored specifically to the individual patient based on the genetic and/or molecular profile of the patient is urgently needed. Among patients scheduled for neoadjuvant chemotherapy, the investigators should differentiate between patients who will be highly effective with neoadjuvant chemotherapy and those who will not, and preferentially select other treatments including radical cystectomy in the patients with high probability of failure to neoadjuvant chemotherapy. However, there is no standard which patients would benefit from neoadjuvant chemotherapy. This study plans to predict treatment response to neoadjuvant chemotherapy in patients with muscle-invasive bladder cancer by analyzing genetic and molecular profiles of tumor tissues obtained through transurethral bladder tumor resection.

ELIGIBILITY:
Inclusion criteria:

* Suspicious of bladder cancer scheduled to have transurethral resection of bladder tumor
* Consent to the provision of their biospecimen.
* Willing to cooperate with this study and comply with the restrictions.
* Voluntarily signed the consent form for participation in the study.
* Age ≥18.

Exclusion criteria:

* Do not agree with this study.
* Vulnerable participants

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Drop-out criteria:
  * Not following treatment schedule (transurethral resection of bladder tumor -> neoadjuvant chemotherapy -> radical cystectomy)
  * Severe side effects during chemotherapy
  * Do not want to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2033-11 (Estimated); Study Completion 2033-11 (Estimated)

PRIMARY OUTCOMES:
Identification of responder to neoadjuvant chemotherapy by genetic and molecular profiles | At the end of 2 cycles of neoadjuvant chemotherapy (each cycle is 14 days (for ddMVAC) / 28 days (for GC))
  Evaluation of the treatment response to neoadjuvant chemotherapy of muscle-invasive bladder cancer patients by imaging (CT and/or MRI) using the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) and correlate with the genetic and molecular profiles of samples (tissue, urine, and blood) analyzed by spatial transcriptomics.

SECONDARY OUTCOMES:
overall survival of bladder cancer patients who have undergone neoadjuvant chemotherapy and radical cystectomy | within 10 years after the neoadjuvant chemotherapy and radical cystectomy
  - Evaluation of the overall survival of bladder cancer patients who have undergone neoadjuvant chemotherapy and radical cystectomy
cancer-specific survival of bladder cancer patients who have undergone neoadjuvant chemotherapy and radical cystectomy | within 10 years after the neoadjuvant chemotherapy and radical cystectomy
  - Evaluation of the cancer-specific survival of bladder cancer patients who have undergone neoadjuvant chemotherapy and radical cystectomy
progression-free survival of bladder cancer patients who have undergone neoadjuvant chemotherapy and radical cystectomy | within 10 years after the neoadjuvant chemotherapy and radical cystectomy
  - Evaluation of the progression-free survival of bladder cancer patients who have undergone neoadjuvant chemotherapy and radical cystectomy
recurrence-free survival of bladder cancer patients who have undergone neoadjuvant chemotherapy and radical cystectomy | within 10 years after the neoadjuvant chemotherapy and radical cystectomy
  - Evaluation of the recurrence-free survival of bladder cancer patients who have undergone neoadjuvant chemotherapy and radical cystectomy

CONTACTS AND LOCATIONS:
Overall Officials: Won Sik Ham, Principal Investigator — Department of Urology and Urological Science Institute, Yonsei University College of Medicine Seoul, Republic of Korea
Locations (1):
- Department of Urology and Urological Science Institute, Yonsei University College of Medicine Seoul, Republic of Korea, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No